CLINICAL TRIAL: NCT02079298
Title: Safety of Fluconazole Treatment of Premature and Full-term Newborn Infants - A Study on Interactions by Nonsteroidal Anti Inflammatory Drugs (NSAIDs) With Fluconazole in Respect of Pharmacodynamic Endpoints With Urinary Excretion of Vasoactive Endobiotics
Brief Title: Safety of Fluconazole Treatment of Premature and Full-term Newborn Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anders Rane, MD, PhD, Senior professor (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Anders Rane, MD, PhD, Senior professor, Senior professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EudraCT number: 2013-003611-21
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Ductus Arteriosis, Patent; Bacterial Infections and Mycoses
MeSH Terms: conditions — Bacterial Infections and Mycoses | interventions — Therapeutics; Fluconazole; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Premature newborn infants with Gestational Age 23+0 to 26+6 weeks who are treated only with fluconazole.
  Interventions: Drug: Treatment with fluconazole.
- 2 (Active Comparator): Premature newborn infants with Gestational Age 23+0 to 26+6 weeks who are treated with both fluconazole and Ibuprofen.
  Interventions: Drug: 2. Treatment with both fluconazole and Ibuprofen.
- 3 (Active Comparator): Premature newborn infants with Gestational Age 27+0 to 36+6 who are treated only with ibuprofen.
  Interventions: Drug: 3. Treatment with ibuprofen.
- 4 (Placebo Comparator): Premature newborn infants with Gestational Age 27+0 to 36+6 and fullterm infants who are not treated either with fluconazole or ibuprofen.
  Interventions: Other: 4. No treatment with either fluconazole nor ibuprofen.

INTERVENTIONS:
Drug: Treatment with fluconazole.
  Arms: 1
Drug: 2. Treatment with both fluconazole and Ibuprofen.
  Arms: 2
Drug: 3. Treatment with ibuprofen.
  Arms: 3
Other: 4. No treatment with either fluconazole nor ibuprofen.
  Arms: 4

SUMMARY:
This study will investigate pharmacological interventions between fluconazole and ibuprofen when they are given to premature newborn babys. This in order to find out if the drugs are influencing each other when they are given at the same time. The study is meant to find out if there are reasons to adjust the dose when fluconazole and ibuprofen are given together.

DETAILED DESCRIPTION:
To evaluate the effect of fluconazole and/or ibuprofen on the urinary excretion of two vasoactive arachidonic acid products, thromboxane A2 (TXA2) and prostacycline (PGI2), in newborn infants treated with one or both of these drugs because of fungal infection prophylaxis and/or patent ductus arteriosis (PDA), respectively, as measurement of the possible interactions between these drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn infants in need of prophylaxis with fluconazole according to clinical routines and/or clinical indication for treatment of Patent Ductus Arteriosis (PDA), or newborn infants who are not treated with either fluconazole or ibuprofen according to the following study groups:

   1.1 Premature newborn infants with Gestational Age 23+0 to 26+6 weeks who are treated only with fluconazole.

   1.2 Premature newborn infants with Gestational Age 23+0 to 26+6 weeks who are treated with both fluconazole and Ibuprofen.

   1.3 Premature newborn infants with Gestational Age 27+0 to 36+6 who are treated only with ibuprofen.

   1.4 Premature newborn infants with Gestational Age 27+0 to 36+6 and fullterm infants who are not treated either with fluconazole or ibuprofen.
2. Parents that are in command of the Swedish language and capable of understanding the study plan
3. Informed written parental consent

Exclusion Criteria:

1. Infants who need treatment with other drugs that are metabolised by enzyme Cytochrome (CYP2C9) (such as phenytoin, sulphamethoxazole, fluvastatin, sildenafil, losartan, irbesartan, torsemide, tienilic acid), or any other enzyme involved in the metabolism of fluconazole and or NSAIDs, or treatment with drugs that interact with NSAIDs at the cyclooxygenase level, or interact with the vasal effects of the metabolic products of the cyclooxygenase.
2. Infants without possibility to conceive the objectives and implications of the study in the opinion of the investigator.

Ages: 23 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Urinary concentrations of prostacycline (PGI2) and thromboxane A2 (TxA2) measured in picogram/milliliter. | 5 days
  To evaluate the effect of fluconazole and/or ibuprofen on the urinary excretion of two vasoactive arachidonic acid products, thromboxane A2 (TXA2) and prostacycline (PGI2), in newborn infants treated with one or both of these drugs for fungal infection prophylaxis and/or patent ductus arteriosis (PDA), respectively.

SECONDARY OUTCOMES:
Concentration of thromboxane A2 (TXA2) and prostacycline (PGI2) in relation to genetic variation of the enzymes of the Cytochrome (P4502C) family. | 5 days
  To evaluate if genetic variability in the enzyme Cytochrome (P4502C) influence the urinary excretion of two vasoactive arachidonic acid products: thromboxane A2 (TXA2) and prostacycline (PGI2) in newborn infants treated with fluconazole and/or ibuprofen.
Number of and type of Adverse Drug Reactions | 5 days
  To evaluate safety of fluconazole and ibuprofen given separately or in combination to newborn infants with clinical indication for treatment with these drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rane, Prof. MD, Study Director — Karolinska Institutet
Locations (1):
- Neonatal Intensive Care Unit, Karolinska University Hopsital, Stockholm, Sweden